CLINICAL TRIAL: NCT07279948
Title: A Single-arm Observational Study to Characterize the Demographic, Clinical Features and Outcomes of a Brazilian Cohort of Patients With Lung Cancer.
Acronym: LUSIP
Status: Not yet recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D133FR00225
Record Dates: First submitted 2025-12-01; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-11

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A single-arm observational study to characterize the demographic, clinical features and outcomes of a Brazilian cohort of patients with lung cancer.

DETAILED DESCRIPTION:
Main hypothesis: The tomographic screening for lung cancer in a population with a high prevalence of granulomatous disease could leads to an increase in the proportion of false-positive cases resulting in unnecessary medical procedures, which represents a waste of resources and a risk for patients.

Main objective: To assess whether the percentage of false-positive cases with indication of biopsy after lung cancer screening with low-dose CT in high-risk smokers in a population with a high prevalence of granulomatous disease will be within the expected range according to other studies in the literature.

As there is robust evidence of the effectiveness of screening in reducing mortality from lung cancer, we expect the project to bring benefits to patients treated for image-detected lung cancer in the project, with reduced staging and a shorter time between diagnosis and treatment. Therefore , although the focus is on the safety of screening, the project will also monitor the cancer detection rate, which is a surrogate endpoint of effectiveness.

ELIGIBILITY:
Inclusion Criteria:

In order, to be eligible for the study, patients must fulfill all the following inclusion criteria:

* Age between ≥50 and ≤80 years.
* Be a current smoker or have quit 15 years ago or less.
* Have participated or are currently participating in smoking cessation program.
* Lifetime smoking exposure equal to or greater than 20 pack-year.
* Provided signed informed consent (ICF)

Exclusion Criteria:

* In order, to be exclude for the study, patients must at least one of the following exclusion criteria:

  * Contraindications to the screening examination: (claustrophobic or weighing more than 130 kgs).
  * Inability to climb 3 stair steps non-stop (36 steps).
  * Disabling dyspnea
  * Symptomatic (with signs and symptoms suspicious of breast cancer lung, namely):

    * pleuritic chest pain
    * rapidly progressive dyspnea of recent onset
    * hemoptysis
    * unexplained hoarseness, lasting more than 1 month.
    * bone pain
    * supraclavicular lymphadenopathy or cervical lymphadenopathy persistent
    * unexplained weight loss of 5% or more of weight in less than 6 months
    * Previous history of malignant neoplasm (excluding non-melanoma skin cancer) diagnosed less than 10 years before the date of the interview;
    * Patients with diagnostic of severe psychiatric disease
    * Immunosuppressed by illness or drugs.
    * Subjected to anterior lung resection even when determined due to an etiology other than malignant neoplasia.
    * Person with a serious terminal illness that contraindicates curative lung surgery.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The population of this study will be adult patients, both sexes, a high-risk smoker selected from a population with a high prevalence of granulomatous disease. The smokers at high risk for developing lung cancer, in a population with a high prevalence of granulomatous disease made up of SUS users registered in the Smoking Cessation Program in the Municipality of Rio de Janeiro, Brazil.
Sampling Method: Non-Probability Sample
Enrollment: 477 (Estimated)
Dates: Start 2026-02-24 (Estimated); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
• Proportion of negative cases on screening according to the Lung-RADS classification. | Last 10 years
  Tomographic screening for lung cancer in a population with a high prevalence of granulomatous disease may increase the proportion of false-positive cases, leading to unnecessary medical procedures, resource waste, and patient risk. This epidemiological scenario may also result in an increase in cases classified as benign or probably benign in screening.
• Proportion of false-positives. | Last 10 years
  Tomographic screening for lung cancer in a population with a high prevalence of granulomatous disease may increase the proportion of false-positive cases, leading to unnecessary medical procedures, resource waste, and patient risk. This epidemiological scenario may also result in an increase in cases classified as benign or probably benign in screening.

SECONDARY OUTCOMES:
• Cancer detection rate. | last 10 years
  Not Applicable (N/A). The findings of each outcome will be compared with results published in the scientific literature.
• Willingness to be screened (ie, proportion of eligible patients actually signing up for the study) | Last 10 years
  Not Applicable (N/A). The findings of each outcome will be compared with results published in the scientific literature.
• Percentage of adherence to screening - calculated by dividing the number of individuals screened with LDCT (numerator) by the number of eligible individuals invited to screen (denominator). | Last 10 years
  Not Applicable (N/A). The findings of each outcome will be compared with results published in the scientific literature.
• Percentage of adherence to follow-up. | Last 10 years
  Not Applicable (N/A). The findings of each outcome will be compared with results published in the scientific literature.
• Prevalence of granulomatous disease in screening positive cases | Last 10 years
  Not Applicable (N/A). The findings of each outcome will be compared with results published in the scientific literature.
• Prevalence of incidental findings. | Last 10 years
  Not Applicable (N/A). The findings of each outcome will be compared with results published in the scientific literature.
• Prevalence of clinically relevant incidental findings that required follow-up. | Last 10 years
  Not Applicable (N/A). The findings of each outcome will be compared with results published in the scientific literature.

OTHER OUTCOMES:
• Willingness to be screened (ie, proportion of eligible patients actually signing up for the study) | Last 10 years
  Not Applicable (N/A). The findings of each outcome will be compared with results published in the scientific literature.
• Percentage of adherence to screening - calculated by dividing the number of individuals screened with LDCT (numerator) by the number of eligible individuals invited to screen (denominator). | Last 10 years
  Not Applicable (N/A). The findings of each outcome will be compared with results published in the scientific literature.

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Rio de Janeiro, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/